CLINICAL TRIAL: NCT06042829
Title: Impact of Covid-19 Aerosol Box On Intubation Success Rate and Intubation Time
Brief Title: Impact of Covid-19 Aerosol Box On Intubation Success Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HTM-2020-006
Record Dates: First submitted 2021-06-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Intubation; Difficult or Failed
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubation with aerosol box (Experimental): Aerosol box group where patient will be intubated using aerosol box
  Interventions: Device: Intubation using aerosol box
- Intubation without Aerosol box (Active Comparator): Without aerosol box group whereby patients will be intubated without aerosol box.
  Interventions: Device: Intubation without aerosol box

INTERVENTIONS:
Device: Intubation using aerosol box — Intubation time and ease of intubation using aerosol box
  Arms: Intubation with aerosol box
Device: Intubation without aerosol box — Intubation time and ease of intubation without aerosol box
  Arms: Intubation without Aerosol box

SUMMARY:
The safety of novel medical device must be assessed before being implemented into clinical practice. In the case of aerosol box, one of the safety features concerned includes its impact on intubation and how it affect the probability of efficient intubation in order to avoid risk of hypoxia to patient. As the barrier box is newly invented, there have been limited studies published.

This study aims to compare intubation success rate between intubation with and without aerosol box in real patients, which will determine the chances of efficient intubation and reflect the safety features of the aerosol box.

DETAILED DESCRIPTION:
General Objective To determine whether intubation performed using aerosol box will have a lower chance of success as compared to intubation without using the box.

Specific Objectives

1. To determine whether intubation with aerosol box will require more time for successful intubation as compared to intubation without the box.
2. To compare the ease of intubation and determine whether intubation using aerosol box will require additional airway manipulation as compared to intubation without using the box.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. American Society of Anesthesiologist (ASA) I or II patients
3. Tested negative for COVID-19 prior to surgery
4. Patient scheduled for elective surgery under general anaesthesia

Exclusion Criteria:

1. Claustrophobia
2. Difficult airway features
3. Body mass index (BMI) of more than 35 kg/m2
4. Body habitus not physically fit into the aerosol box.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Tracheal intubation time | 1 year
  Time taken from the laryngoscope blade passes through front incisors, followed by endotracheal intubation being inserted into trachea, and until the first upstroke of the capnograph trace visible as proof of successful tracheal intubation (the measurement is measured in seconds)

SECONDARY OUTCOMES:
Ease of tracheal intubation | 1 year
  Based on scale of tracheal intubation difficulty. The scale is called Intubation Difficulty Scale. Intubation difficulty scale is a numerical score of total intubation difficulty and is based on seven parameters known to be associated with difficult intubation. The seven parameters are number of attempts, number of intubators, number of alternative techniques, Cormack-Lehane laryngoscopy grades, requirement of lifting force of laryngoscopy, application of laryngeal pressure, and mobility of vocal cords. The score will be summed. The degree of difficulty will be categorized into easy (IDS score of 0), slight difficulty (IDS of 1-4) and moderate to major difficulty (IDS of 5 and more) according to the total score. The higher score is associated with a higher prevalence of difficult intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Najwa Mohd Noor Dr, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia